CLINICAL TRIAL: NCT04626336
Title: Post-operative Hernias After Radical Cystectomy : Incidence and Risks Factors
Brief Title: Post-operative Hernias After Radical Cystectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0604
Record Dates: First submitted 2020-11-02; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Evisceration; Traumatic; Hernia
Keywords: Median hernia; Parastomal hernia; Cystectomy
MeSH Terms: conditions — Hernia | interventions — Cystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who undergo a cystectomy: Patients who undergo a cystectomy for cancer or not, since 2010 to 2020
  Interventions: Procedure: Cystectomy

INTERVENTIONS:
Procedure: Cystectomy — Cystectomy

SUMMARY:
Post-operative hernias after cystectomy are frequent (our review of the literature with meta-analysis found an incidence of evisceration at 5%, median eventrations at 8% and peristomal hernias at 14%). These represent a non-negligible and partially morbidity. avoidable, subject to proper assessment of personal and surgical risk factors

ELIGIBILITY:
Inclusion criteria:

* having undergone a cystectomy (for cancer or not),
* with or without reconstruction, between 01/01/2010 and 12/31/2020

Exclusion criteria:

- refusing to participate

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo cystectomy for cancer or not at the CHU de Montpellier, Nîmes and the Beau Soleil clinic
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2010-01-30 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Type of post-operative hernias | 1 day
  Type of post-operative hernias : evisceration, median hernia, parastomal hernia
Define risk factors Type of risks factors | 1 day
  Define risk factors: sex, BMI, diabetes, ASA, duration surgery, delay, postoperative biology

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Aujoulat, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC